CLINICAL TRIAL: NCT06358248
Title: Standardized Physician-modified Fenestrated Endograft Registry
Acronym: SPHERE
Status: Recruiting | Type: Observational
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Michele Piazza, Principal Investigator, University Hospital Padova
Other Study IDs: SPHERE
Record Dates: First submitted 2024-04-07; First posted 2024-04-10 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Aortic Aneurysm, Thoracoabdominal; Aortic Diseases
Keywords: Aortic Aneurysm; Thoracoabdominal Aneurysm; Endovascular aortic repair
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal; Aortic Diseases; Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients treated: All patients treated with 4-fen PMEG endograft
  Interventions: Device: Physician-modification of Valiant Captivia Endograft (Medtronic, Minneapolis, MN-USA).

INTERVENTIONS:
Device: Physician-modification of Valiant Captivia Endograft (Medtronic, Minneapolis, MN-USA). — On a sterile back-table a Valiant Captivia thoracic graft is deployed. A dotted line is drawn to mark the graft anterior 0° degree, and fabric holes are performed with cautery in the desired position. The fenestrations need to be 6x6 mm for the renals and 8x8 mm for superior mesenteric artery (SMA) and celiac trunk (CT), and are reinforced with the tip of a 0.018 guidewire through a continuous 5-0 locking suture.
  A posterior constraining wire is created to reduce the diameter of the graft by 20-30%, in order to allow rotation during the deployment phase. The four "8" markers on the top of the graft are carefully removed with a scalpel; one of these is modified as an "S" and re-sutured on the anterior aspect at 0 degree position, with a 5-0 prolene continuous suture. This "S" marker will allow anteroposterior graft orientation. Finally, the graft is re-sheathed and deployed.

SUMMARY:
Multicenter retrospective study including all consecutive patients treated by PMEG using a standard modification technique of Valiant Captivia (Medtronic, Minneapolis, MN-USA).

DETAILED DESCRIPTION:
INTRODUCTION

Abdominal aortic aneurysms (AAA) without an adequate proximal neck length for safe sealing and fixation with a standard EVAR may benefit from complex endovascular repair. The most common are short neck AAA, juxta/para-renal AAA, and type IV thoracoabdominal aneurysm (TAAA), where incorporation of renal and visceral vessels is required to obtain an adequate proximal sealing. Several endovascular options are available, with the most effective being represented by incorporation of target vessels by custom-made or off-the-shelf fenestrated/branched endografts.

Custom-made devices have shown excellent early and long-term outcomes, but due to manufacturing time (up to three months), they can be used only for elective cases. In urgent cases, readily available off-the-shelf devices can be used, but their anatomical feasibility is not exhaustive, and may require long segment of aortic coverage above the celiac trunk. Parallel aortic grafts with chimneys or periscopes have been proposed as a timely alternative; however, gutter endoleaks and lack of proximal sealing are serious concerns for these techniques, especially for those cases where more than two target vessels need to be incorporated.

In patients presenting with large aneurysm, symptomatic, or requiring urgent repair, the use of physician-modified endograft (PMEG) represents a valid option. It allows for a rapid customization of a standard abdominal or thoracic device with the creation of fenestrations, scallops or branches, based on patient aneurysm anatomical extent and target vessel position.

However, these techniques demand high level of skills and experience; a recent review showed also that in the literature there is an extreme variability on indication to treatment, type of aneurysm and extension, type of graft, and method of modification, thus limiting the possibility to adequately analyze outcomes or drive comparison between different techniques.

Here the investigators describe an initial experience on safety and feasibility of a standardized approach with PMEG, based on specific anatomical selection criteria, measurement method and a standard technique of modification, using the Valiant Captivia (Medtronic, Minneapolis, MN-USA) thoracic endograft.

BACKGROUND AND PRELIMINARY DATA

The vast majority of the literature on PMEG is based on the Cook platform. Recently Chait et al. reported the long term outcomes of more than 150 Cook PMEGs, with excellent results in terms of early mortality, freedom from aortic-related mortality, and target instability, especially for complex AAA compared to TAAA.

There is only a single experience using Valiant Captivia PMEG Valiant in the version without free-flow. In this experience the authors reported 18 cases; after complete unsheathing, the graft was introduced in a sterile aortic 3D model for precise fenestration allocation and then re-sheathed. The investigators think that leaving the graft on its device may reduce the risk of infection, reducing manipulation and contact with other materials, as the the printed aortic model. The other two case reports using the Valiant platform for the treatment of the paravisceral segment are from Gibello et al., that used a Valiant Navion graft, and Joseph et al., that applied mini-cuff-augmented fenestration using Valiant Captivia.

STANDARDIZED DEVICE MODIFICATION

The graft is modified on a sterile back-table in a hybrid operating room, while the patient is prepared for general anesthesia. A Valiant Captivia thoracic graft with free-flow (either with tubular or tapered shape) is fully deployed without releasing the free-flow, that is maintained retained on its tip. After that, a vertical dotted line is drawn to mark the graft anterior 0° degree, and fabric holes are performed with ophthalmologic cautery in the desired position, taking care of not having graft struts within the fenestrations. The fenestrations need to be nicely round, ideally 6x6 mm for the renals and 8x8 mm for superior mesenteric artery (SMA) and celiac trunk (CT), and are reinforced with the tip of a 0.018 guidewire (V-18, Boston Scientific, Marlborough, Massachusetts-USA) through a continuous 5-0 non-adsorbable locking suture (Ti-cron, Medtronic, Minneapolis, Minnesota-USA).

A posterior constraining wire is created to temporarily reduce the diameter of the graft by 20-30%, in order to allow partial rotation during the deployment phase. The back of a 0.018'' guidewire is routed on the posterior aspect of the graft passing within the external suture of the struts, thus not requiring fabric puncture; the prolene used to reduce the diameter are tied around the stent struts and subsequently looped to the posterior wire. The four "8" markers on the top of the graft are carefully removed with a scalpel; one of these is modified as an "S" and re-sutured on the anterior aspect at 0 degree position, with a 5-0 prolene continuous suture. This "S" marker will allow anteroposterior graft orientation. Finally, the graft is re-sheathed with help of vessel loop.

FOLLOW-UP

A postoperative CTA is required within 30 days. Further follow-up follow-up is left to each center, but ideally includes imaging follow-up at 6, 12, 24 months and yearly thereafter.

ELIGIBILITY:
INCLUSION CRITERIA

* Complex AAA (including short-neck AAA, JRAA, PRAA, extent IV TAAA)
* Haemodynamic stability
* Anatomical feasibility is based on the presence of a proximal aortic neck above the mid celiac trunk of ≥25 mm in length and between 18 mm and 35 mm in diameter; the neck needs to be "healthy" with no parietal calcifications or thrombus with a cylindrical shape. The visceral aorta is required to be no larger than 40 mm in maximum diameter.

EXCLUSION CRITERIA

* Extent I-III TAAA
* Hemorrhagic shock

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent e PMEG with 4-fenestration procedure for the treatment of a short neck AAA, juxta/para-renal AAA, and type IV thoracoabdominal aneurysm (TAAA).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2033-10-01 (Estimated)

PRIMARY OUTCOMES:
Technical success | Intra-operative
  Number of participants who underwent a successful deployment of the endograft and stenting of the 4 visceral vessels
Freedom from target vessel instability | 5 years
  Number of participants who experience any occlusion, endoleak, aneurysm rupture, stent restenosis needing a re-intervention
Freedom from endograft instability | 5 years
  Number of participants who show absence of endoleak, aneurysm rupture, endograft migration

SECONDARY OUTCOMES:
Early (30-days) Major Adverse Event (MAE) | 5 years
  Any early (30-days) Major Adverse Event
Aneurysm sac dynamics | 5 years
  Number of participants who experience aneurysm sac diameter change during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Michele Piazza, MD, Principal Investigator — University Hospital Padova
Locations (1):
- Vascular and Endovascular Clinic - Padova University, Padua, Italy